CLINICAL TRIAL: NCT04292366
Title: Optimising Colorectal Cancer Screening Participation -A Randomised Controlled Trial of Invitation Procedures
Brief Title: Optimising Colorectal Cancer Screening Participation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: participationCRC2020
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Neoplasms
Keywords: mass screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention arm I (Experimental): pre-notification approximately ten days prior to intervention, invitation and one reminder (three-staged intervention)
  Interventions: Procedure: Invitation procedure
- Intervention arm II (Experimental): invitation, one reminder after 45 days and a second reminder three months after invitation (three-staged invitation procedure)
  Interventions: Procedure: Invitation procedure
- Intervention arm III (Experimental): pre-notification, invitation, reminder after 45 days and reminder after three months (four-staged invitation procedure)
  Interventions: Procedure: Invitation procedure
- Control group (Active Comparator): invitation and one reminder after 45 days (usual care)
  Interventions: Procedure: Invitation procedure

INTERVENTIONS:
Procedure: Invitation procedure — Optimised invitation procedures in an organised colorectal cancer screening programme

SUMMARY:
The aim of this study is to demonstrate the effectiveness of three and four-staged invitation procedures compared to two-staged procedures by combining pre-notifications and reminders. The RCT will be nested into the Danish colorectal cancer screening programme in the Central Denmark Region including men and women aged 50-74 years. Participants will consecutively be randomized into four arms in a 1:1 ratio. Intervention arm 1 will receive a pre-notification approximately ten days prior to intervention, invitation and one reminder (three-staged intervention), Intervention arm 2 will receive invitation, one reminder after 45 days and a second reminder three months after invitation (three-staged invitation procedure), Intervention arm 3 will receive pre-notification, invitation, reminder after 45 days and reminder after three months (four-staged invitation procedure). Finally, the forth arm will be a control group receiving usual care which invitation and one reminder 45 days after invitation (two-staged invitation procedure). Both pre-notifications and reminders are sent using digital mail.

The main out-come will be participation within 6 months after invitation.

ELIGIBILITY:
Inclusion Criteria:

* Invited for colorectal cancer screening

Exclusion Criteria:

-

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60000 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Number of residents participating in colorectal cancer screening | Within six months after invitaiton
  Number of residents participating in colorectal cancer screening in each of the four arms

CONTACTS AND LOCATIONS:
Overall Officials: Berit Andersen, Professor, Study Director — Randers Regional Hospital
Locations (1):
- Randers Regional Hospital, Randers, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen MB, Hedelund M, Flander L, Andersen B. The impact of pre-notifications and reminders on participation in colorectal cancer screening - A randomised controlled trial. Prev Med. 2022 Nov;164:107229. doi: 10.1016/j.ypmed.2022.107229. Epub 2022 Aug 31. PMID 36057390